CLINICAL TRIAL: NCT03851406
Title: Phase I/II Randomized Cross-over Study of Hypertonic Saline on Airway Inflammatory Response to Inhaled Wood Smoke
Brief Title: Woodsmoke Particulate + Hypertonic Saline
Acronym: Smokeysal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18-1895
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-02

CONDITIONS: Airway Inflammation

STUDY DESIGN:
Intervention Model Description: To determine the efficacy of nebulized 5% hypertonic saline (HS) (v. no treatment) in mitigating wood smoke particulate (WSP)-induced neutrophilic airway inflammation, assessed via sputum %polymorphonuclear leukocytes (PMNs), in healthy adults 4 hours post WSP exposure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 5% Hypertonic Saline, then No Inhaled Treatment (Active Comparator): Participants will receive 5% Hypertonic Saline following WSP exposure. After a 2-week washout period, participants will receive no treatment following WSP exposure.
  Interventions: Device: 5% Hypertonic Saline; Other: No treatment
- No Inhaled Treatment, then 5% Hypertonic Saline (Active Comparator): Participants will receive no inhaled treatment following WSP exposure. After a 2-week washout period, participants will receive 5% Hypertonic Saline following WSP exposure.
  Interventions: Device: 5% Hypertonic Saline; Other: No treatment

INTERVENTIONS:
Device: 5% Hypertonic Saline — Immediately following exit from the wood smoke chamber, participants will inhale 15 mL of 5% Hypertonic Saline for 15 minutes delivered by Pari neb with a coached cough maneuver.
Other: No treatment — No inhaled treatment will be provided immediately following exit from the wood smoke chamber.

SUMMARY:
Deployment of military personnel has been associated with increased respiratory illness likely due, in part, to inhalation of unusual particulate matter (PM), such as from burn pits. Inflammation is a key initial response to inhaled particulates. The investigator has developed a protocol using inhaled wood smoke particles (WSP) as a way to study PM-induced airway inflammation. Exposure to wood smoke particles causes symptoms, even in healthy people, such as eye irritation, cough, shortness of breath, and increased mucous production. The purpose of this research study is to see if a single treatment of inhaled hypertonic saline (HS) can diminish this PM-induced airway inflammation by rapidly clearing the WSP inhaled particles from airway surfaces. The exposure will be 500 ug/m³ of WSP for 2 hours, with intermittent exercise on a bicycle and rest. The wood is burned in a typical wood stove and piped into the chamber.

DETAILED DESCRIPTION:
Military deployment is associated with exposure to novel particulate matter (PM), such as from burn pits, aeroallergens, and increased cigarette consumption. War fighters exposed to these inhalational exposures exhibit immediate and chronic respiratory morbidity. For example, military service personnel surveyed in both the Republic of Korea (ROK) and Kabul, Afghanistan reported a general increase in respiratory morbidity, including asthma and chronic bronchitis, associated with their deployment. Air contaminants in the ROK were characterized by elevated levels of both PM 0.5-2.5 and PM 2.5-10. Similarly, exposures in Kabul were characterized by multiple airborne PM exposures, including those from burn pits. Burn pit PM includes metals, bioaerosols, organic by-products, and biomass combustion particles. These findings indicate that inhaled PM is a likely cause of respiratory morbidity in the field.

Inflammation is a key initial response to inhaled particulates. Wood smoke particles (WSP) serve as a model agent to study PM-induced bronchitis. WSP inhalation generates reactive oxidant (and nitrosative) species which cause local injury of airway epithelial cells and release of damage-associated molecular patterns (DAMPs) that activate toll-like receptors (TLR) and interleukin 1 (IL-1)-mediated innate immune responses by resident airway macrophages. Contamination of PM with bioaerosols, which contain lipopolysaccharide (LPS), also activates innate immune responses through toll-like receptor 4 (TLR4) activation of resident airway macrophages. These complementary processes result in recruitment of neutrophils (PMN), which mediate luminal airway inflammation with release of toxic mediators such as neutrophil elastase and myeloperoxidase that promote acute and chronic bronchitis.

Therefore, mitigation of PM-induced airway neutrophilic inflammation should be a key focus in order to reduce the respiratory morbidity of military personnel. The investigators have studied a number of pro-inflammatory inhaled agents, such as nebulized LPS, ozone (O3), and WSP, as models of acute neutrophilic bronchitis against which to test a number of therapeutic agents. To this effect, the investigators have reported that inhaled fluticasone inhibits O3-induced and LPS-induced neutrophilic inflammation, and that parenteral anakinra and oral gamma-tocopherol inhibit neutrophilic responses to inhaled LPS. In addition to agents with inherent anti-inflammatory and anti-oxidant properties, rapid clearance of inhaled particles from airway surfaces is a complementary approach to reduce PM-induced airway inflammation. This can be assessed through the measurement of mucociliary clearance (MCC).

MCC is dependent on airway secretory cells and submucosal glands that produce a mucin-rich fluid layer on the airway surface and ciliated cells that hydrate and propel mucus out of the lung and into the upper airway. Rates of MCC are dependent on ciliary beat frequency, hydration, and the rheologic properties of mucus. In vitro studies have demonstrated that HS, through an osmotic effect on airway surfaces, improved hydration and mucus rheologic properties, and accelerated mucus transport rates. In addition, the data over the last 30 years has shown that inhaled hypertonic saline (HS) plus cough is the most effective method for acutely clearing the bronchial airways of inhaled, deposited particles. The combined effect is greater than either HS or cough alone. In the studies of asthmatics, the investigators examined the ability of a single HS treatment with a coached cough maneuver to acutely clear radiolabeled Tc99m sulfur colloid particles from airways following LPS exposure. Following HS inhalation and cough clearance maneuvers developed to recover sputum samples for analysis, the investigators observed a rapid clearance of >50% of the inhaled radiolabelled particles. The investigators hypothesize that if other pro-inflammatory particles (PMs, burn pit particles) were cleared similarly via HS-induced acceleration of MCC shortly after exposure, there would be reductions in acute PM-induced inflammation. Thus, in this study, the investigators will assess the effectiveness of inhaled 5% HS, a dose well tolerated by asthmatics at baseline and after inhaled LPS/allergen challenges for sputum induction, in mitigating WSP-induced airway neutrophilic inflammation in healthy volunteers. Normal saline 0.9% (NS) is not going to be used as a placebo treatment in this study, as inhalation of NS itself impacts the rheologic properties of mucus and MCC and thus would not be a suitable placebo. The investigators will, therefore, compare treatment with 5% HS to no receiving no treatment following WSP exposure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years, inclusive, of both genders
* Negative pregnancy test for females who are not s/p hysterectomy with oophorectomy
* No history of episodic wheezing, chest tightness, or shortness of breath consistent with asthma, or physician-diagnosed asthma.
* forced expiratory volume at one second (FEV1) of at least 80% of predicted and FEV1/forced vital capacity (FVC) ratio of >0.70.
* Oxygen saturation of >93%
* Ability to provide an induced sputum sample.
* Subject must demonstrate a >10% increase in sputum %PMNs 6 hours following inhaled WSP exposure, when compared to baseline sputum (to be completed in a separate protocol #15-1775).
* Proof of vaccination to SARS-CoV-2 based on public health guidelines at time of inclusion

Exclusion Criteria:

* Clinical contraindications:
* Any chronic medical condition considered by the PI as a contraindication to the exposure study including significant cardiovascular disease, diabetes, chronic renal disease, chronic thyroid disease, history of chronic infections/immunodeficiency.
* Viral upper respiratory tract infection within 4 weeks of challenge.
* Any acute infection requiring antibiotics within 4 weeks of exposure or fever of unknown origin within 4 weeks of challenge.
* Abnormal physical findings at the baseline visit, including but not limited to abnormalities on auscultation, temperature of 37.8° C, Systolic BP > 150mm Hg or < 85 mm Hg; or Diastolic BP > 90 mm Hg or < 50 mm Hg, or pulse oximetry saturation reading less than 93%.
* Physician diagnosis of asthma
* If there is a history of allergic rhinitis, subjects must be asymptomatic of allergic rhinitis at the time of study enrollment.
* Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.
* Medications which may impact the results of the WSP exposure, interfere with any other medications potentially used in the study (to include steroids, beta antagonists, non-steroidal anti-inflammatory agents)
* Cigarette smoking > 1 pack per month
* Unwillingness to use reliable contraception if sexually active (IUD, birth control pills/patch, condoms).
* Use of immunosuppressive or anticoagulant medications including routine use of NSAIDS. Oral contraceptives are acceptable, as are antidepressants and other medications may be permitted if, in the opinion of the investigator, the medication will not interfere with the study procedures or compromise safety and if the dosage has been stable for 1 month.
* Orthopedic injuries or impediments that would preclude bicycle or treadmill exercise.
* Inability to avoid NSAIDS, Multivitamins, Vitamin C or E or herbal supplements.
* Allergy/sensitivity to study drugs or their formulations
* Positive COVID-19 test in the past 90 days.
* Pregnant/lactating women and children (< 18 years as this is age of majority in North Carolina) will also be excluded since the risks associated with WSP exposure to the fetus or child, respectively, are unknown and cannot be justified for this non-therapeutic protocol. Individuals over 45 years of age will not be included due to the increased possibility of co-morbidities and need for prohibited medications.
* Inability or unwillingness of a participant to give written informed consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terry Noah, M.D, Principal Investigator — UNC Chapel Hill
Locations (1):
- Center for Environmental Medicine, Asthma and Lung Biology at UNC Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pugh MJ, Jaramillo CA, Leung KW, Faverio P, Fleming N, Mortensen E, Amuan ME, Wang CP, Eapen B, Restrepo M, Morris MJ. Increasing Prevalence of Chronic Lung Disease in Veterans of the Wars in Iraq and Afghanistan. Mil Med. 2016 May;181(5):476-81. doi: 10.7205/MILMED-D-15-00035. PMID 27136656
- [Background] Korzeniewski K, Nitsch-Osuch A, Konior M, Lass A. Respiratory tract infections in the military environment. Respir Physiol Neurobiol. 2015 Apr;209:76-80. doi: 10.1016/j.resp.2014.09.016. Epub 2014 Sep 30. PMID 25278277
- [Background] Baird CP. Review of the Institute of Medicine report: long-term health consequences of exposure to burn pits in Iraq and Afghanistan. US Army Med Dep J. 2012 Jul-Sep:43-7. No abstract available. PMID 22815164
- [Background] Gomez JC, Yamada M, Martin JR, Dang H, Brickey WJ, Bergmeier W, Dinauer MC, Doerschuk CM. Mechanisms of interferon-gamma production by neutrophils and its function during Streptococcus pneumoniae pneumonia. Am J Respir Cell Mol Biol. 2015 Mar;52(3):349-64. doi: 10.1165/rcmb.2013-0316OC. PMID 25100610
- [Background] Barth SK, Dursa EK, Bossarte R, Schneiderman A. Lifetime Prevalence of Respiratory Diseases and Exposures Among Veterans of Operation Enduring Freedom and Operation Iraqi Freedom Veterans: Results From the National Health Study for a New Generation of U.S. Veterans. J Occup Environ Med. 2016 Dec;58(12):1175-1180. doi: 10.1097/JOM.0000000000000885. PMID 27930474
- [Background] Szema AM. Occupational Lung Diseases among Soldiers Deployed to Iraq and Afghanistan. Occup Med Health Aff. 2013;1:10.4172/2329-6879.1000117. doi: 10.4172/2329-6879.1000117. PMID 24443711
- [Background] Morris MJ, Lucero PF, Zanders TB, Zacher LL. Diagnosis and management of chronic lung disease in deployed military personnel. Ther Adv Respir Dis. 2013 Aug;7(4):235-45. doi: 10.1177/1753465813481022. Epub 2013 Mar 7. PMID 23470637
- [Background] Auerbach A, Hernandez ML. The effect of environmental oxidative stress on airway inflammation. Curr Opin Allergy Clin Immunol. 2012 Apr;12(2):133-9. doi: 10.1097/ACI.0b013e32835113d6. PMID 22306553
- [Background] Alexis NE, Brickey WJ, Lay JC, Wang Y, Roubey RA, Ting JP, Peden DB. Development of an inhaled endotoxin challenge protocol for characterizing evoked cell surface phenotype and genomic responses of airway cells in allergic individuals. Ann Allergy Asthma Immunol. 2008 Mar;100(3):206-15. doi: 10.1016/S1081-1206(10)60444-9. PMID 18426139
- [Background] Hernandez ML, Harris B, Lay JC, Bromberg PA, Diaz-Sanchez D, Devlin RB, Kleeberger SR, Alexis NE, Peden DB. Comparative airway inflammatory response of normal volunteers to ozone and lipopolysaccharide challenge. Inhal Toxicol. 2010 Jul;22(8):648-56. doi: 10.3109/08958371003610966. PMID 20540623
- [Background] Hernandez M, Brickey WJ, Alexis NE, Fry RC, Rager JE, Zhou B, Ting JP, Zhou H, Peden DB. Airway cells from atopic asthmatic patients exposed to ozone display an enhanced innate immune gene profile. J Allergy Clin Immunol. 2012 Jan;129(1):259-61.e1-2. doi: 10.1016/j.jaci.2011.11.007. PMID 22196529
- [Background] Alexis NE, Peden DB. Blunting airway eosinophilic inflammation results in a decreased airway neutrophil response to inhaled LPS in patients with atopic asthma: a role for CD14. J Allergy Clin Immunol. 2001 Oct;108(4):577-80. doi: 10.1067/mai.2001.118511. PMID 11590384
- [Background] Hernandez ML, Mills K, Almond M, Todoric K, Aleman MM, Zhang H, Zhou H, Peden DB. IL-1 receptor antagonist reduces endotoxin-induced airway inflammation in healthy volunteers. J Allergy Clin Immunol. 2015 Feb;135(2):379-85. doi: 10.1016/j.jaci.2014.07.039. Epub 2014 Sep 5. PMID 25195169
- [Background] Hernandez ML, Wagner JG, Kala A, Mills K, Wells HB, Alexis NE, Lay JC, Jiang Q, Zhang H, Zhou H, Peden DB. Vitamin E, gamma-tocopherol, reduces airway neutrophil recruitment after inhaled endotoxin challenge in rats and in healthy volunteers. Free Radic Biol Med. 2013 Jul;60:56-62. doi: 10.1016/j.freeradbiomed.2013.02.001. Epub 2013 Feb 9. PMID 23402870
- [Background] Burbank AJ, Duran CG, Pan Y, Burns P, Jones S, Jiang Q, Yang C, Jenkins S, Wells H, Alexis N, Kesimer M, Bennett WD, Zhou H, Peden DB, Hernandez ML. Gamma tocopherol-enriched supplement reduces sputum eosinophilia and endotoxin-induced sputum neutrophilia in volunteers with asthma. J Allergy Clin Immunol. 2018 Apr;141(4):1231-1238.e1. doi: 10.1016/j.jaci.2017.06.029. Epub 2017 Jul 20. PMID 28736267
- [Background] Alexis NE, Hu SC, Zeman K, Alter T, Bennett WD. Induced sputum derives from the central airways: confirmation using a radiolabeled aerosol bolus delivery technique. Am J Respir Crit Care Med. 2001 Nov 15;164(10 Pt 1):1964-70. doi: 10.1164/ajrccm.164.10.2104051. PMID 11734453
- [Background] Alexis NE, Lay JC, Zeman KL, Geiser M, Kapp N, Bennett WD. In vivo particle uptake by airway macrophages in healthy volunteers. Am J Respir Cell Mol Biol. 2006 Mar;34(3):305-13. doi: 10.1165/rcmb.2005-0373OC. Epub 2005 Nov 4. PMID 16272458
- [Background] Sood N, Bennett WD, Zeman K, Brown J, Foy C, Boucher RC, Knowles MR. Increasing concentration of inhaled saline with or without amiloride: effect on mucociliary clearance in normal subjects. Am J Respir Crit Care Med. 2003 Jan 15;167(2):158-63. doi: 10.1164/rccm.200204-293OC. Epub 2002 Oct 31. PMID 12411282
- [Background] Alexis NE, Bennett W, Peden DB. Safety and benefits of inhaled hypertonic saline following airway challenges with endotoxin and allergen in asthmatics. J Asthma. 2017 Nov;54(9):957-960. doi: 10.1080/02770903.2016.1278019. Epub 2017 Jan 17. PMID 28095128
- [Background] Ghio AJ, Soukup JM, Case M, Dailey LA, Richards J, Berntsen J, Devlin RB, Stone S, Rappold A. Exposure to wood smoke particles produces inflammation in healthy volunteers. Occup Environ Med. 2012 Mar;69(3):170-5. doi: 10.1136/oem.2011.065276. Epub 2011 Jun 30. PMID 21719562
- [Background] Esther CR Jr, Lazaar AL, Bordonali E, Qaqish B, Boucher RC. Elevated airway purines in COPD. Chest. 2011 Oct;140(4):954-960. doi: 10.1378/chest.10-2471. Epub 2011 Mar 31. PMID 21454402
- [Background] Jones B, and Kenward, M.G. . Design and analysis of cross-over trials. Third ed: CRC Press; 2015.
- [Background] Alexis NE, Zhou H, Lay JC, Harris B, Hernandez ML, Lu TS, Bromberg PA, Diaz-Sanchez D, Devlin RB, Kleeberger SR, Peden DB. The glutathione-S-transferase Mu 1 null genotype modulates ozone-induced airway inflammation in human subjects. J Allergy Clin Immunol. 2009 Dec;124(6):1222-1228.e5. doi: 10.1016/j.jaci.2009.07.036. PMID 19796798

RESULTS

PARTICIPANT FLOW:
Groups:
- 5% Hypertonic Saline, Then No Inhaled Treatment: Participants received 5% Hypertonic Saline following WSP exposure. After a 2-week washout period, participants received no treatment following wood smoke particles (WSP) exposure.
  5% Hypertonic Saline: Immediately following exit from the wood smoke chamber, participants will inhale 15 mL of 5% Hypertonic Saline for 15 minutes delivered by Pari neb with a coached cough maneuver.
  No treatment: No inhaled treatment will be provided immediately following exit from the wood smoke chamber.
- No Inhaled Treatment, Then 5% Hypertonic Saline: Participants received no inhaled treatment following WSP exposure. After a 2-week washout period, participants received 5% Hypertonic Saline following WSP exposure.
  5% Hypertonic Saline: Immediately following exit from the wood smoke chamber, participants will inhale 15 mL of 5% Hypertonic Saline for 15 minutes delivered by Pari neb with a coached cough maneuver.
  No treatment: No inhaled treatment will be provided immediately following exit from the wood smoke chamber.
Period: First Intervention
Arm/Group | 5% Hypertonic Saline, Then No Inhaled Treatment | No Inhaled Treatment, Then 5% Hypertonic Saline
Started | 4 | 5
Received Intervention | 4 | 3
Received no Intervention | 0 | 2
Completed | 4 | 3
Not Completed | 0 | 2
Period: Washout (2 Weeks)
Arm/Group | 5% Hypertonic Saline, Then No Inhaled Treatment | No Inhaled Treatment, Then 5% Hypertonic Saline
Started | 4 | 3
Completed | 4 | 2
Not Completed | 0 | 1
Period: Second Intervention
Arm/Group | 5% Hypertonic Saline, Then No Inhaled Treatment | No Inhaled Treatment, Then 5% Hypertonic Saline
Started | 3 (One participant did not return for the second intervention.) | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5% Hypertonic Saline, Then No Inhaled Treatment | No Inhaled Treatment, Then 5% Hypertonic Saline | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 4 Hours in Sputum Percent Neutrophils
Description: Change in sputum percent neutrophils from baseline to 4 hours post WSP exposure
Time Frame: Baseline, 4 hours post WSP exposure
Population: An attempt was made to analyze samples for all participants; although some samples had an inadequate cell differential slide. Data are reported for all samples that yielded data for each endpoint and at each time.
Measure: Median (Inter-Quartile Range); unit: percent neutrophils
Groups:
- 5% Hypertonic Saline: Participants received 5% Hypertonic Saline following WSP exposure.
  5% Hypertonic Saline: Immediately following exit from the wood smoke chamber, participants will inhale 15 mL of 5% Hypertonic Saline for 15 minutes delivered by Pari neb with a coached cough maneuver.
- No Inhaled Treatment: Participants received no inhaled treatment following WSP exposure.
  No treatment: No inhaled treatment will be provided immediately following exit from the wood smoke chamber.
Arm/Group | 5% Hypertonic Saline | No Inhaled Treatment
Number analyzed (Participants) | 5 | 5
percent neutrophils | -0.04 [-12 to 12] | -0.5 [-3.7 to 1.4]
Statistical Analysis 1: Comparison: 5% Hypertonic Saline vs No Inhaled Treatment; Test type: Other; p > 0.99, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05

2. Primary Outcome: Change From Baseline to 24 Hours in Sputum Percent Neutrophils
Description: Change in sputum percent neutrophils from baseline to 24 hours post WSP exposure
Time Frame: Baseline, 24 hours post WSP exposure
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent neutrophils
Arm/Group | 5% Hypertonic Saline | No Inhaled Treatment
Number analyzed (Participants) | 6 | 5
percent neutrophils | 17 [-0.25 to 30] | 29 [1.5 to 36]
Statistical Analysis 1: Comparison: 5% Hypertonic Saline vs No Inhaled Treatment; Test type: Other; p > 0.99, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05

3. Secondary Outcome: Change in Number of Sputum Neutrophils
Description: Neutrophil numbers/mg compared at 4 and 24 hours post WSP exposure with respect to Baseline.
Time Frame: Baseline, 4 and 24 hours post WSP exposure
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Neutrophils/mg
Arm/Group | 5% Hypertonic Saline | No Inhaled Treatment
Number analyzed (Participants) | 6 | 5
Neutrophils/mg
  4 hours post WSP exposure: number analyzed (Participants) | 5 | 5
  4 hours post WSP exposure | 0.40 [-6.9 to 203] | 19 [-41 to 70]
  24 hours post WSP exposure | 9.5 [-261 to 174] | 79 [16 to 148]
Statistical Analysis 1: Comparison: 5% Hypertonic Saline vs No Inhaled Treatment; 4 hours post WSP exposure; Test type: Other; p > 0.99, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05
Statistical Analysis 2: Comparison: 5% Hypertonic Saline vs No Inhaled Treatment; 24 hours post WSP exposure; Test type: Other; p > 0.99, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05

4. Secondary Outcome: Change in Number of Sputum Eosinophils
Description: Eosinophil numbers/mg compared at 4 and 24 hours post WSP exposure with respect to Baseline.
Time Frame: Baseline, 4 and 24 hours post WSP exposure
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Eosinophils/mg
Arm/Group | 5% Hypertonic Saline | No Inhaled Treatment
Number analyzed (Participants) | 6 | 5
Eosinophils/mg
  4 hours post WSP exposure | 0 [-1.3 to 28] | 0 [-0.32 to 0.42]
  24 hours post WSP exposure | -0.10 [-1.4 to 0.74] | 0.45 [-0.18 to 3.3]
Statistical Analysis 1: Comparison: 5% Hypertonic Saline vs No Inhaled Treatment; 4 hours post WSP exposure; Test type: Other; p = 0.38, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05
Statistical Analysis 2: Comparison: 5% Hypertonic Saline vs No Inhaled Treatment; 24 hours post WSP exposure; Test type: Other; p = 0.38, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05

5. Secondary Outcome: Change in Percent Sputum Eosinophils
Description: Percent eosinophils compared at 4 and 24 hours post WSP exposure with respect to Baseline.
Time Frame: Baseline, 4 and 24 hours post WSP exposure
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent eosinophils
Arm/Group | 5% Hypertonic Saline | No Inhaled Treatment
Number analyzed (Participants) | 6 | 5
percent eosinophils
  4 hours post WSP exposure | 0.33 [0.00 to 0.89] | 0.00 [-0.24 to 0.11]
  24 hours post WSP exposure | 0.00 [-0.23 to 0.12] | 0.00 [-0.11 to 13.00]
Statistical Analysis 1: Comparison: 5% Hypertonic Saline vs No Inhaled Treatment; 4 hours post WSP exposure; Test type: Other; p = 0.25, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05
Statistical Analysis 2: Comparison: 5% Hypertonic Saline vs No Inhaled Treatment; 24 hours post WSP exposure; Test type: Other; p = 0.63, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05

6. Secondary Outcome: Change in Interleukin-1b
Description: Interleukin-1β via the Mesoscale platform (pg/mL) compared at 4 and 24 hours post-WSP exposure with respect to Baseline.
Time Frame: Baseline, 4 and 24 hours post WSP exposure
Population: An attempt was made to analyze samples for all participants; although some samples had an insufficient sample quantity. Data are reported for all samples that yielded data for each endpoint and at each time.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | 5% Hypertonic Saline | No Inhaled Treatment
Number analyzed (Participants) | 6 | 5
pg/mL
  4 hours post WSP exposure | 0.95 [-7.7 to 3.8] | -2.5 [-5.5 to -0.23]
  24 hours post WSP exposure | 0.41 [-6.3 to 7.8] | -0.58 [-7.8 to 1.6]
Statistical Analysis 1: Comparison: 5% Hypertonic Saline vs No Inhaled Treatment; 4 hours post WSP exposure; Test type: Other; p = 0.88, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05
Statistical Analysis 2: Comparison: 5% Hypertonic Saline vs No Inhaled Treatment; 24 hours post WSP exposure; Test type: Other; p > 0.99, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05

7. Secondary Outcome: Change in Interleukin-6
Description: Interleukin-6 via Mesoscale platform (pg/mL) compared at 4 and 24 hours post WSP exposure with respect to Baseline.
Time Frame: Baseline, 4 and 24 hours post WSP exposure
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | 5% Hypertonic Saline | No Inhaled Treatment
Number analyzed (Participants) | 6 | 5
pg/mL
  4 hours post WSP exposure | 0.94 [-2.1 to 4.4] | -1.2 [-3.4 to 1.4]
  24 hours post WSP exposure | 0.73 [-1.2 to 35] | -1.9 [-2.2 to 5.7]
Statistical Analysis 1: Comparison: 5% Hypertonic Saline vs No Inhaled Treatment; 4 hours post WSP exposure; Test type: Other; p = 0.88, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05
Statistical Analysis 2: Comparison: 5% Hypertonic Saline vs No Inhaled Treatment; 24 hours post WSP exposure; Test type: Other; p = 0.25, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05

8. Secondary Outcome: Change in Interleukin-8
Description: Interleukin-8 via Mesoscale platform (pg/mL) compared at 4 and 24 hours post WSP exposure with respect to Baseline.
Time Frame: Baseline, 4 and 24 hours post WSP exposure
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | 5% Hypertonic Saline | No Inhaled Treatment
Number analyzed (Participants) | 6 | 5
pg/mL
  4 hours post WSP exposure | -37 [-232 to 1027] | -138 [-209 to 95]
  24 hours post WSP exposure | 65 [-55 to 177] | 82 [-322 to 437]
Statistical Analysis 1: Comparison: 5% Hypertonic Saline vs No Inhaled Treatment; 4 hours post WSP exposure; Test type: Other; p > 0.99, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05
Statistical Analysis 2: Comparison: 5% Hypertonic Saline vs No Inhaled Treatment; 24 hours post WSP exposure; Test type: Other; p > 0.99, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05

9. Secondary Outcome: Change in Tumor Necrosis Factor Alpha
Description: Tumor Necrosis Factor Alpha via Mesoscale platform (pg/mL) compared at 4 and 24 hours post WSP exposure with respect to Baseline.
Time Frame: Baseline, 4 and 24 hours post WSP exposure
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | 5% Hypertonic Saline | No Inhaled Treatment
Number analyzed (Participants) | 6 | 5
pg/mL
  4 hours post WSP exposure | 0.00 [-3.60 to 0.81] | -0.35 [-0.39 to -0.05]
  24 hours post WSP exposure | 0.05 [-0.10 to 11.00] | 0.22 [-0.38 to 0.37]
Statistical Analysis 1: Comparison: 5% Hypertonic Saline vs No Inhaled Treatment; 4 hours post WSP exposure; Test type: Other; p = 0.75, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05
Statistical Analysis 2: Comparison: 5% Hypertonic Saline vs No Inhaled Treatment; 24 hours post WSP exposure; Test type: Other; p = 0.38, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05

10. Other Pre Specified Outcome: Mucociliary Clearance (MCC)
Description: 4 hours post WSP exposure, the MCC is done. A whole lung region of interest (ROI) bordering the right lung is used to estimate (by computer analysis) whole lung retention of inhaled radiolabeled particles. Labeled particle counts are measured over a 2 hour period to determine the fraction of initial particle counts remaining. From this data, the investigators will determine the percentage of labeled particles cleared from the lung during the 2 hour observation period.
Time Frame: 4 hours post WSP exposure]
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through final follow-up visit which occurred one week after the final wood smoke exposure, up to 3 months.
Arm/Group | 5% Hypertonic Saline | No Inhaled Treatment
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5% Hypertonic Saline (N=6) | No Inhaled Treatment (N=6)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nose bleed (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT03851406/Prot_SAP_001.pdf
  • Informed Consent Form (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT03851406/ICF_000.pdf